CLINICAL TRIAL: NCT04255472
Title: Effectiveness of the WHO Caregivers Skills Training (CST) Program for Children With Developmental Disorders and Delays in Rural Community Settings in Pakistan: An Individual Randomized Controlled Trial (RCT)
Brief Title: Effectiveness of the WHO Caregivers Skills Training Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Human Development Research Foundation, Pakistan (Other)
Collaborators: World Health Organization (Other); University of Liverpool (Other); Benazir Bhutto Hospital, Rawalpindi (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WHO CST-RCT
Record Dates: First submitted 2019-09-14; First posted 2020-02-05 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Autism Spectrum Disorder; Development Delay; Developmental Disorder; Language Delay; Behavioral Problem; Emotional Problem; Maternal Distress
MeSH Terms: conditions — Autism Spectrum Disorder; Learning Disabilities; Developmental Disabilities; Language Development Disorders; Problem Behavior | interventions — galactosylceramide sulfotransferase; Therapeutics

STUDY DESIGN:
Intervention Model Description: Two arm, single blind individual randomized controlled trial (RCT)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors will be blind to the allocations status of participants. To ensure blinding, participants will be instructed to not disclose their allocation during assessment.
  Fidelity of masking will be ensured by having assessors guess the allocation status of participants at the end of assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WHO caregiver skills training program (Experimental): Strategies to support children's communication skills by learning to engage in play activities and daily home routines activities with their caregivers.
  Interventions: Behavioral: WHO Caregiver skills training (CST) program
- Treatment as usual (TAU) (Experimental): TAU in primary healthcare centers for childhood developmental disorders and delays usually consists of no treatment, or a range of alternate treatment regimes, such as multi-vitamin syrups and tablets.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: WHO Caregiver skills training (CST) program — Caregivers are provided with tangible strategies to appropriately respond to their children's emotional regulation, engagement, and communication. Further, the program focuses on helping caregivers to develop their children's communication and adaptive skills while reducing challenging behavior by focusing on identifying the function of the behavior and learning to teach developmentally appropriate replacement skills. The WHO CST program includes nine group sessions delivered at a community venue (e.g., BHU, school, home) and three home visits: the first at entry prior to session 1, the second after session 4, and the third after the final group session. Training for program facilitators will be included prior to the delivery of the intervention.
  Arms: WHO caregiver skills training program
Behavioral: Treatment as usual — WHO CST will be compared with TAU. TAU in primary healthcare centers for childhood developmental disorders and delays usually consists of no treatment, or a range of alternate treatment regimes, such as multi-vitamin syrups and tablets. Evidence-based mental health care is currently not available in primary healthcare centers. A complete record of services availed by the trial participants at tertiary mental healthcare center will be maintained by using an adapted Client Services Receipt Inventory (CSRI) for children with developmental disorders and delays at baseline and end point.
  Arms: Treatment as usual (TAU)

SUMMARY:
Background: Increasing prevalence rates of developmental disorders (DDs) including Autism Spectrum Disorders (ASD) and intellectual disability are a public health priority particularly in Low and Middle Income countries (LIMC) and are included in the World Health Organization (WHO) mhGAP program. However, existing mental health care facilities and resources are insufficient in most low resource settings to cater for this increasing demand. To address this situation, Caregiver Skills Training (CST) program for children with developmental disorders and delays has been developed by the WHO to bridge the treatment gap in low resource settings.

Objective: The objective of this study is to evaluate the effectiveness of the WHO CST program plus treatment as usual (TAU) vs. TAU to improve caregiver-child interaction in children with developmental disorders and delays, when implemented by non-specialist health care facilitators in a low-resource rural community settings of Rawalpindi, Pakistan.

Methods: A two arm, single blind individual randomized controlled trial (RCT) will be carried out with 160 caregiver-child dyads with development disorders and delays in community settings of Rawalpindi, Pakistan. 160 caregiver-child dyads will be individually randomized on 1:1 allocation ratio into intervention (n=80) and control (n=80) arms. Participants in the intervention arm will receive 3-hours group training sessions of WHO CST program once every week for 9 weeks and 3 individual home sessions delivered via non-specialist health care facilitator over a duration of 3-months. The primary outcome is improvement in play-based caregiver-child interaction at 9-months post-intervention. The secondary outcomes are improvement in routine home-based caregiver-child interaction, child's social communication skills, adaptive behavior, emotional and behavioral problems and parental health related quality of life. The data on health services utilization will also be collected at 9-months post-intervention. Qualitative process evaluation with a sub-sample of study participants and trainers will be undertaken following the RCT. The study will be completed within an estimated period of 11-months.

Discussion: Outcomes of the study will be the evidence on the effectiveness of WHO CST program to improve caregiver child interaction and improvement in social communication skills, adaptive behaviors of children with developmental disorders and delays in the low resource setting of Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-9 years old, with developmental disorders and delays as screened by TQS
* Screened positive on communication problems as identified by Communication and Symbolic Behavior Scale (CSBS) score <41
* Developmental Disability-Children's Global Assessment Scale (DD-CGAS) score ≥ 51 as assessed by clinician.

Exclusion Criteria:

* Children having epilepsy with seizures in the previous 6 months
* Children with Cerebral Palsy as assessed by the clinician.
* Co-morbid physical and mental conditions in the child that require inpatient hospitalization.
* Significant uncorrected hearing and visual impairment in child or parent.
* Any severe psychiatric or physical illness in primary caregiver requiring inpatient hospitalization.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Play-based caregiver-child interaction | 9-months post-intervention
  The primary outcome will be change in play-based caregiver-child interaction using Joint Engagement Rating Inventory. An observational, video rated tool will be used to rate caregivers-child's engagement and behavior during play and home routine following a communication play protocol on a 7-point Likert scale The tool has been adapted for coding. caregivers' child interaction in the context of Pakistan. Fifteen-minute video taped caregiver-child interaction will be collected at baseline and at endpoint for families in both arms of the study. Caregivers will be asked to try play based routines (e.g. playing with toys or reading a book) with their child or home routines involving the child (e.g. feeding the child performing domestic chores). The videos will be singly coded by trained assessors.

SECONDARY OUTCOMES:
Adaptive functioning behaviors | At baseline, 9-weeks and 9-months post-intervention follow-up.
  Vineland Adaptive Behavior Scales (VABS) will be used to measure adaptive behaviors. VABS will be used to measure child's functioning in the area of communication, daily living skills, socialization and motor skills. The VABS contains 5 domains each with 2-3 subdomains. The main domains are Communication, Daily Living Skills, Socialization, Motor Skills, and Maladaptive Behavior (optional). There are five general categories of answers for each item. These are "Usually Performs", "Sometimes Perform", "Never Performs", Never had the opportunity to perform" and "Don't know or never observed the child to perform".
Child emotional and behavioral problems | At baseline, 9-weeks and 9-months post-intervention follow-up.
  Child emotional and behavioral problems will be measured through Child Behavior Checklist (CBCL). It consists of 113 questions, scored on a three-point Likert scale (0=absent, 1= occurs sometimes, 2=occurs often). CBCL is made up of eight syndrome scales: anxious/depressed, depressed, somatic complaints, social problems, thought problems, attention problems, rule-breaking behavior, and aggressive behavior.
Parental health related quality of life | At baseline, 9-weeks and 9-months post-intervention follow-up.
  Parental health related quality of life will be measured by Pediatric Quality of Life (PedsQL) Family impact module. It is a 36 items impact module scale that consisting of 6 sub-scales measuring parent self-reported functioning. These subscales measure physical functioning, emotional functioning, social functioning, daily activities and family relationships. Items are rated on a 5-point Likert scale (0 = never to 4= almost always) and add up to 100 score, where higher scores indicate better Health Related Quality of Life.
Health services utilization | At baseline and 9-months post-intervention follow-up.
  The cost of health services utilization from the time proceeding assessment will be assessed with the adapted Client Services Receipt Inventory (CSRI). It has been adapted to use for the families of children with developmental disorders and delays. It measures the utilization of various health and social care services including time and opportunity losses by the families in the care of their child with developmental disorder and delay.
Communication and Symbolic Behavior | Screening, 9-weeks & 9-months post-intervention follow-up.
  Communication and Symbolic Behavior Scale will be used as a screening tool to identify children with delay in social communication, expressive speech/language, and symbolic functioning, as well as a secondary outcome measures to determine the impact of intervention overtime. CSBS measures 7 language predictors: emotion and eye gaze, communication, gestures, sounds, words, understanding, and object use. CSBS caregiver questionnaire consists of 41 items divided into seven clusters which make three composites i.e. social composite, speech composite and symbolic composite. Items are rated on 3-point Likert scale: "Not Yet/Rarely", "Sometimes" and "Often/Usually".

CONTACTS AND LOCATIONS:
Overall Officials: Syed Usman Hamdani, PhD, Principal Investigator — Human Development Research Foundation, Pakistan
Locations (1):
- Human Development Research Foundation, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] mhGAP Intervention Guide for Mental, Neurological and Substance Use Disorders in Non-Specialized Health Settings: Mental Health Gap Action Programme (mhGAP). Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK138690/ PMID 23741783
- [Background] Chisholm D, Knapp MR, Knudsen HC, Amaddeo F, Gaite L, van Wijngaarden B. Client Socio-Demographic and Service Receipt Inventory--European Version: development of an instrument for international research. EPSILON Study 5. European Psychiatric Services: Inputs Linked to Outcome Domains and Needs. Br J Psychiatry Suppl. 2000;(39):s28-33. doi: 10.1192/bjp.177.39.s28. PMID 10945075
- [Background] Wetherby, A.M. and B.M. Prizant, Communication and symbolic behavior scales (CSBS). 2003: Brookes Publishing Company.
- [Background] Sparrow SS, Cicchetti DV. Diagnostic uses of the Vineland Adaptive Behavior Scales. J Pediatr Psychol. 1985 Jun;10(2):215-25. doi: 10.1093/jpepsy/10.2.215. No abstract available. PMID 4020603
- [Background] Varni JW, Seid M, Rode CA. The PedsQL: measurement model for the pediatric quality of life inventory. Med Care. 1999 Feb;37(2):126-39. doi: 10.1097/00005650-199902000-00003. PMID 10024117